CLINICAL TRIAL: NCT03170167
Title: Effectiveness of a Mind-Body and Peer Support Program for Teens Living With Chronic Illness and Their Parents: A Pilot Study
Brief Title: Communitas: A Program for Teens Living With Chronic Illness and Their Families
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Rick Hecht, Research Director of the Osher Center, and Professor of Medicine at UCSF, University of California, San Francisco
Other Study IDs: 13-11679
Record Dates: First submitted 2016-10-18; First posted 2017-05-30 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Chronic Illness
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: This is a pre-post survey study of Communitas, a pre-existing integrative medicine and mind-body skills group visit for adolescents living with chronic illness and their parents. Approximately 50-100 patient enrollees of the Communitas group visits will be recruited to participate in this survey study optionally.
- Parents: This is a pre-post survey study of Communitas, a pre-existing integrative medicine and mind-body skills group visit for adolescents living with chronic illness and their parents. Approximately 50-100 parent enrollees of the Communitas group visits will be recruited to participate in this survey study optionally.

SUMMARY:
The proposed pilot study is an evaluation of Communitas, a mind-body skills group visit and for 12-19 year-olds living with chronic physical illness. The goal of this study is to assess the efficacy and feasibility of these group visits. During 2017-2018, the investigators will recruit 50-100 patient and 50-100 parent enrollees of Communitas to participate in this study. The study will be a pre-post evaluation, without a control group, using validated patient-report assessments at baseline, after completion of the group visits, and 3 months later. The primary outcome variables will be physical and mental wellbeing, stress, mood, resilience, mindfulness, and social support. Paired t tests will be used to assess changes from baseline to immediately post-intervention & 3 months post-intervention. The investigators will also calculate Cohen's d effect sizes, to help them understand the degree to which an effect is present in the population.

DETAILED DESCRIPTION:
The Communitas pilot study is a survey study of Communitas, a pre-existing integrative medicine and mind-body skills group visit for adolescents living with chronic illness and their parents. The goal of this study is to evaluate the preliminary efficacy and feasibility for these group visits. Approximately 50-100 patients and 50-100 parent enrollees of the Communitas group visits will be recruited to participate in this survey study optionally. During the group visits, both the patient and parent groups will learn about and experience various coping, self-care, pain and stress-reduction modalities, participate in group sharing to promote engagement with a diagnosis and provide emotional support, and benefit from facilitated discussions about some of the more practical aspects of living with chronic illness. The group visits will be offered to patients and their parents as clinical service, regardless of enrollment in the survey study, and will be billed to insurance as consult group visit with the pediatrician. The group visits will be held at both the Osher Center for Integrative Medicine and Mission Bay Children's Hospital and will be led by a pediatrician, starting in October 2016. The study will be set up as a pre-post evaluation, without a control group, using patient-report and parent-report qualitative and quantitative assessments at baseline, after completion of the series of group visits, and 3 months later. In addition, some families may be asked if they would like to participate in a videotaped interview before and after the start of the program.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Communitas group visit at the UCSF Osher Center for Integrative Medicine or Mission Bay Children's Hospital.
* Patients enrolled in these group visits are males and females 12-20 years of age and living with a chronic illness.

Exclusion Criteria:

* People who are not enrolled in the Communitas group visit at the UCSF Osher Center for Integrative Medicine or Mission Bay Children's Hospital will be excluded from this survey study.
* The Communitas group consists of a patient group of young people ages 12-20 living with chronic illness, as well as a parent group.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 12-20 year-old pediatric patients who are living with a chronic physical illness and who are enrolled in the Communitas group visit at the UCSF Osher Center for Integrative Medicine or Mission Bay Children's Hospital, along with their willing and available guardian(s).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Physical wellbeing | Change from baseline NIH Promis Global Health instrument summary score at 2 months and at 5 months
  NIH Promis Global Health instrument summary score
Mental wellbeing | Change from baseline NIH Promis Global Health instrument summary score at 2 months and at 5 months
  NIH Promis Global Health instrument summary score
Perceived Stress | Change from baseline Perceived stress scale summary score at 2 months, and at 5 months
  Perceived stress scale summary score
Mood: Tension | Change from baseline Profile of Mood States Tension instrument subscale score at 2 months and at 5 months
  Profile of Mood States Tension instrument subscale score
Resilience | Change from baseline 14-Item Resilience Scale summary score at 2 months and at 5 months
  14-Item Resilience Scale summary score
Social support | Change from baseline Social Support Scale summary score at 2 months, and at 5 months
  Social Support Scale summary score
Mindfulness | Change from baseline Mindful Attention Awareness Scale summary score at 2 months, and at 5 months
  Mindful Attention Awareness Scale summary score
Mood: Anger | Change from baseline Profile of Mood States Anger instrument sub scale score at 2 months, and at 5 months
  Profile of Mood States Anger instrument subscale score
Mood: Depression | Change from baseline Profile of Mood States Depression instrument sub scale score at 2 months, and at 5 months
  Profile of Mood States Depression instrument subscale score
Mood: Fatigue | Change from baseline Profile of Mood States Fatigue instrument sub scale score at 2 months, and at 5 months
  Profile of Mood States Fatigue instrument subscale score

SECONDARY OUTCOMES:
Self-reported adherence, using Medical Outcomes Study General Adherence scale | Change from baseline Medical Outcomes Study General Adherence instrument summary score at 2 months, and at 5 months
  Medical Outcomes Study General Adherence instrument summary score
pain medicine usage in past month | Change from baseline pain medicine usage in past month likert scale at 2 months, and at 5 months
  likert scale
number visits to emergency department in past month | Change from baseline number visits to emergency department in past month at 2 months, and at 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Hecht, MD, Principal Investigator — UCSF Osher Center for Integrative Medicine
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided